CLINICAL TRIAL: NCT06002126
Title: Optimization of Cervical Cancer Screening Among Women Living With HIV in Latin American Countries
Acronym: ULACNet-202
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); H. Lee Moffitt Cancer Center and Research Institute (Other); University of Sao Paulo (Other); Mexican National Institute of Public Health (Other Government); University of California, San Diego (Other); Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-02025683; U54CA242639 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Cervix Cancer; HPV Infection; Cervical High Grade Squamous Intraepithelial Lesion; HIV Infections
Keywords: HPV; cervical cancer screening; women with HIV; DNA methylation; extended HPV genotyping
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cervical cancer screening (single arm) (Experimental): Women will be screened for cervical cancer with HPV testing that provides extended genotyping and DNA quantification. Women will also provide other samples for cervical cancer screening tests. Women will under cervical biopsies.
  Interventions: Diagnostic Test: Xpert HPV; Diagnostic Test: QIAsure Methylation Test

INTERVENTIONS:
Diagnostic Test: Xpert HPV — The Cepheid Xpert HPV Assay (Xpert HPV) is a qualitative, real-time polymerase chain reaction (PCR) assay for the detection of hrHPV DNA. The assay is formatted in a single-use, Xpert HPV test cartridge and is run on the Cepheid Xpert® System, a multi-analyte, random access, molecular-diagnostic platform ranging in capacity from 1 to 80 test processing modules. Importantly, a single hrHPV DNA test can be completed in one hour, permitting same-day screening and diagnosis (e.g. colposcopy) or treatment (e.g. cryotherapy), reducing the potential for loss to follow-up in lower-resource settings. It uses liquid-based cytologic media and yields five separate results or channels: HPV 16, HPV 18/45, HPV 31/33/35/52/58, HPV 51/59, HPV 39/68/56/66 all with a corresponding cycle threshold.
Diagnostic Test: QIAsure Methylation Test — The Qiagen QIAsure assay is a multiplex real-time PCR test that amplifies the methylated promoter regions of the tumor suppressor genes, FAM19A4 and has-mir124-2, as well as a methylation-unspecific fragment of the ACTB reference gene. Hypermethylation of the host genes FAM19A4 and has-mir124-2 has been shown to detect high-grade cervical lesions and cancer.

SUMMARY:
Cervical cancer is a relatively common cancer among women living with human immunodeficiency virus (HIV). This study will test women for human papillomavirus (HPV) infection of the cervix. The main purpose of this study is to determine the best way to test for damaged areas of the cervix. Damaged areas of the cervix should be treated and removed to prevent cancer of the cervix.

Women living with HIV (WLWH) in this study will be seen once, twice or three times in a year. Women will provide several samples related to screening for cervical cancer including a swab of the cervix, a self-collected swab of the vagina and urine. Women will have a detailed examination of the cervix called colposcopy and have a few biopsies, or small pinches of the cervix, to look for areas at risk for turning into cancer. If HPV of the cervix is found but treatment of the cervix is not indicated, women will return in 6 months and in 12 months to repeat these tests. Most women will only need 1 visit. Women found to have damaged areas of the cervix at risk for turning into cancer will be referred for treatment.

This protocol will compare different tests to understand the best test to identify women at risk for cervical cancer.

DETAILED DESCRIPTION:
The overall goal of this research is to develop a point of care hrHPV test and molecular testing that optimizes specificity to detect high-grade squamous intraepithelial lesions (HSIL) (namely cervical intraepithelial neoplasia grade 2 or worse, CIN 2+) in WLWH in Latin America while maintaining high test sensitivity. To accomplish this goal, we propose to conduct a trial that optimizes cervical screening by modifying the cycle threshold/genotype interpretation of Xpert HPV assay output. In a secondary manner, we will also evaluate whether triage with host DNA methylation improves the specificity of Xpert alone.

The hypotheses for this protocol includes:

• The Xpert HPV test can be optimized for HSIL detection (CIN2+) in WLWH to significantly improve test specificity, when compared to unmodified test output using manufacturer guidelines.

To evaluate this hypothesis, we will enroll 1000 women aged 25-65 years living with HIV who are undergoing routine cervical cancer screening. These individuals will be recruited from affiliated clinical sites of the Instituto Nacional de Salud Pública in Cuernavaca, Mexico and Universidade de São Paulo in São Paulo, Brazil. Participants will provide a first void urine sample and will be instructed how to self-collect a vaginal swab. An oral gargle specimen will be collected for HPV testing, host DNA methylation, and Epstein-Bar Virus (EBV) co-infection. They will receive a baseline questionnaire about risk factors for HPV and cervical cancer, and provide blood specimens for cluster of differentiation 4/8 (CD4/CD8) count, plasma viral load, as well as future DNA methylation of biological aging and circulating tumor HPV DNA (ctHPVDNA) analysis, and stored sera. Next, a provider will collect an anal swab. Then the participant will undergo a speculum exam, and a provider will collect a cervical cytobroom sample for cytology and HPV testing followed by a swab for stored specimens. Then at least two cervical biopsies will be obtained.

Material from one provider-collected cervical swab will undergo cervical cytology assessment using Bethesda Criteria. Cervical histology results from the collected biopsies will be interpretated according to the Lower Anogenital Squamous Terminology (LAST). HSIL will be defined as CIN 2 with diffuse p16 staining, CIN 2-3, or CIN 3. Women diagnosed with HSIL will be treated according to local standards. The local histology result will be used for the management of participants. Any lesions suspicious for invasive cancer will be referred to the appropriate specialist. Women with HSIL on cytology, but no HSIL on histology will be treated according to the local standard. The management options include repeat colposcopy, endocervical curettage, or a diagnostic loop electro-excision procedure. Similarly, women with a Type 3 transformation zone should have endocervical curettage and be managed according to local standards. After local pathology review, all histology specimens will be shipped centrally for Histology Endpoint Adjudication; these adjudicated histology results will be used for reporting research findings. Discordance between the local and central pathology review will be adjudicated with a second central pathologist. The final histology result will be sent back to the local site and provided to the participant and their providers. Women found to have vulvar, vaginal or perianal lesions suspicious for HSIL will be referred for appropriate evaluation.

The self-collected vaginal swab and material from the provider-collected cytobroom sample will be tested for HPV using Xpert HPV. Xpert testing of self- and provider-collected samples will be conducted locally (at the point of care) in Brazil and Mexico. Remaining material from the vaginal and cervical samples will be shipped to Dr. Villa's lab in Brazil to allow for Qiagen' methylation testing of any WLWH with hrHPV detected. Residual samples, as well as the collected urine, will be stored in Dr. Villa's lab for future studies. In addition, an optional collection of anal canal and a cervical swab will occur in those that specifically provided consent. These specimens will be stored for future medical research and will not be analyzed as part of this study.

Women with hrHPV detected on a provider-collected cervical sample using a locally available and approved test, but who were negative for HSIL as determined by cervical biopsy, will be asked to return for a follow-up study visit at 6-month to receive the same procedures described above (with the exception of blood draws). If at the 6-month follow-up visit WLWH continue to have detection of hrHPV, but are HSIL-negative by biopsy, they will be asked to return for an additional follow-up study visit 6 months later (12-months post-baseline) to receive the same procedures (with blood draws). We estimate that approximately 40% of the population will have hrHPV detected and may need to return for a follow-up visit; and 7% will be HSIL+ and referred for treatment.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infection, as documented by 1) any FDA approved, licensed HIV rapid test performed in conjunction with screening (oral immunoblot, ELISA, test kit, and confirmed by Western blot or other approved test), OR 2) a physician's written record that documents HIV infection with supporting information on the participant's relevant medical history and/or current management of HIV infection, OR 3) documentation of a prescription of an approved antiretroviral regimen by either possession of pill bottles or packages with prescriber's name or ARVs dispensed from an HIV clinical treatment program with two participant identifiers affixed to the bottles or packages.
* Female.
* Aged 25 to 65.
* Ability to understand and the willingness to sign a written informed consent document by the participant or by the legal representative(s) of the participant.

Exclusion Criteria

* History of cervical, vulvar, vaginal, perianal, anal cancer or oral cancer.
* Have undergone cervical cancer screening in the last 6 months.
* Have undergone cervical HSIL treatment in the past year.
* Have a history of hysterectomy with removal of the cervix.
* Have never had sexual intercourse (oral or genital or anal).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (including opportunistic infections of Acquired Immunodeficiency Syndrome-AIDS and/or genitourinary infections), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to the lack of safety data of performing colposcopy during pregnancy.
* Any other medical condition or social situation that would put the participant, the study staff, or the study outcomes at risk, as determined by the site investigators.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cervical HSIL or invasive cancer on histology at baseline | Baseline
  Diagnosis of cervical HSIL (defined as CIN 2 with p16 staining, CIN 2-3, or CIN3) or squamous cell carcinoma from histology of cervical biopsies.

SECONDARY OUTCOMES:
Number of participants with hrHPV at baseline who are found to have cervical HSIL or invasive cancer on histology at Months 6 or 12. | Month 6 or Month 12
  Development of cervical HSIL at the Month 6 or Month 12 visit in WLWH that had detection of hrHPV in cervical or vaginal specimens at the baseline or Month 6 visit.
  Only those subjects that had detection of hrHPV in cervical or vaginal specimens at the baseline or Month 6 visit will be included in the count.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Ellsworth, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- University of São Paulo, São Paulo, Brazil
- National Institute of Public Health, Mexico, Cuernavaca, Morelos, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months post-publication of the primary manuscript through the duration of the NIH award (U54242639).
Access Criteria: Researchers who provide a methodologically sound proposal for use of the data that is approved by the study investigators and the sponsor.
  The research must be broadly consistent with that of ULACNet.
  Researchers may submit a request to the study principal investigator (Grant Ellsworth, gre9006@med.cornell.edu) to request details of request format.